CLINICAL TRIAL: NCT05714007
Title: The Effects of Ferric Derisomaltose on Postoperative Anemia in Patients Undergoing Spinal Deformity Surgery: A Prospective Randomized Controlled Study
Brief Title: The Effects of Ferric Derisomaltose on Postoperative Anemia in Spinal Deformity Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Pharmacosmos A/S (Industry)
Responsible Party: Principal Investigator, Weiyun Chen, Principal Investigator, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PUMCH-Fe
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-02

CONDITIONS: Perioperative Anemia; Surgery; Spinal Deformity; Adult
Keywords: spinal deformity surgery; perioperative anemia; ferric derisomaltose; adult
MeSH Terms: interventions — ferric derisomaltose; ferrous succinate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Iron to be administered as intravenous ferric derisomaltose:
  Where Hb (hemoglobin) ≥100 g/L, dosage according to body weight is as follows:
  Body weight <50 kg: 500mg; Body weight 50 to <70 kg: 1000 mg; Body weight ≥70 kg: 1500 mg.
  Where Hb <100 g/L, dosage according to body weight is as follows:
  Body weight <50 kg: 500mg; Body weight 50 to <70 kg: 1500mg; Body weight ≥70 kg: 2000 mg.
  The maximial dose should not exceed 20mg/kg body weight, rounded off to the nearest 100mg
  Interventions: Drug: Ferric derisomaltose
- Control group (Active Comparator): Iron to be administered as oral ferrous succinate:
  1 tablet (100 mg) tid (three times daily), starting on the first postoperative day and continuing for 4 weeks.
  Interventions: Drug: Ferrous succinate

INTERVENTIONS:
Drug: Ferric derisomaltose — Single intravenous dose ferric derisomaltose
  Other Names: MONOFER®
  Arms: Treatment group
Drug: Ferrous succinate — Daily oral dose of 100 mg iron (ferrous succinate) tid postoperatively
  Arms: Control group

SUMMARY:
The prognosis of patients undergoing spinal deformity surgery is often compromised by perioperative anemia due to iron deficiency. The aim of this randomized, controlled trial was to evaluate whether postoperative ferric derisomaltose intravenous injection may improve anemia and prognosis in patients undergoing spinal deformity surgery comparing with oral iron. Participants will be randomly assigned to the treatment group (intravenous ferric derisomaltose) and the control group (oral iron). Changes in hemoglobin concentration, percentage of anemia correction, changes in iron indicators, patient quality of life, and incidence of adverse events will be analyzed to evaluate the efficacy and safety of iron isomaltoside infusion.

DETAILED DESCRIPTION:
Iron deficiency is a common cause of perioperative anemia in patients undergoing spinal deformity surgery. Anemia may lead to increased postoperative complications and mortalities, prolonged hospital stays, deteriorated physical function, and severely affect the quality of life.

Oral iron has been widely recommended to treat perioperative anemia. However, the pro-inflammatory cytokines (such as IL-6 (Interleukin-6), TNF-a (Tumor necrosis factor-α)) produced by the inflammatory state after surgery can lead to an increase in hepcidin, which greatly affects the absorption of oral iron. Compared to oral iron, intravenous iron can circumvent the effects of decreased iron absorption in the gastrointestinal tract due to the postoperative inflammatory state and achieve faster and more effective iron supplementation. At present, intravenous iron supplements are mainly second-generation products, including iron sucrose and ferric gluconate. However, the unstable molecular structure of second-generation iron supplements may cause oxidative stress, which limits its administration in large doses.

Compared with traditional intravenous iron, the third-generation iron preparations allow more iron (1000 mg (milligram) or more, no more than 20 mg/kg (kilogram)) to be infused within a short period of time (15-60 minutes), improving patient compliance, reducing costs and complications caused by multiple infusions, and is promising to improve anemia more rapidly. Ferric derisomaltose, as the only third-generation iron currently available in China market, has showed its value in treating anemia in joint replacement surgeries. However, the effectiveness of postoperative intravenous ferric derisomaltose in spinal deformity surgery remains uncertain. Therefore, we designed this prospective randomized trial to evaluate whether intravenous ferric derisomaltose may improve anemia and prognosis in patients undergoing spinal deformity surgery compared with oral iron.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years
2. Received spinal deformity surgery
3. 70 g/L ≤ Hb ≤ 110 g/L at POD1, or Hb at POD1 showed a decrease of

   ≥20 g/L compared with baseline
4. Informed consent was obtained voluntarily

Exclusion Criteria

1. Women who are pregnant, breastfeeding, or planning to become pregnant.
2. known serious hypersensitivity to other parenteral iron products
3. Non-iron deficiency anemia (e.g., hemolytic anemia)
4. Decompensated liver insufficiency
5. Coexisting active infection
6. Drug abuse, including but not limited to opioids, amphetamines, methamphetamine, ketamine, etc.
7. Other conditions that the investigator considers inappropriate for participation (e.g. deafness, Parkinson's disease, communication disorders, etc.)
8. Participation in another clinical trial within three months prior to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin concentration | At 14 days
  Change in hemoglobin concentrations from POD(postoperative day)1 to POD14

SECONDARY OUTCOMES:
Change in hemoglobin concentration | At 5 days
  Change in hemoglobin concentrations from POD1 to POD5
Change in hemoglobin concentration | At 35 days
  Change in hemoglobin concentrations from POD1 to POD35
Correction of anemia | At 5 days
  The percentage of effective correction of anemia (elevation of Hb >20g/L or Hb ≥120g/L) at POD5
Correction of anemia | At 14 days
  The percentage of effective correction of anemia (elevation of Hb >20g/L or Hb ≥120g/L) at POD14
Correction of anemia | At 35 days
  The percentage of effective correction of anemia (elevation of Hb >20g/L or Hb ≥120g/L) at POD35
Change in serum iron | At 5 days
  Change in serum iron from POD1 to POD5
Change in serum iron | At 14 days
  Change in serum iron from POD1 to POD14
Change in serum iron | At 35 days
  Change in serum iron from POD1 to POD35
Change in ferritin | At 5 days
  Change in ferritin from POD1 to POD5
Change in ferritin | At 14 days
  Change in ferritin from POD1 to POD14
Change in ferritin | At 35 days
  Change in ferritin from POD1 to POD35
Change in transferrin saturation | At 5 days
  Change in transferrin saturation from POD1 to POD5
Change in transferrin saturation | At 14 days
  Change in transferrin saturation from POD1 to POD14
Change in transferrin saturation | At 35 days
  Change in transferrin saturation from POD1 to POD35
Change in soluble transferrin receptor | At 5 days
  Change in soluble transferrin receptor from POD1 to POD5
Change in soluble transferrin receptor | At 14 days
  Change in soluble transferrin receptor from POD1 to POD14
Change in soluble transferrin receptor | At 35 days
  Change in soluble transferrin receptor from POD1 to POD35
EQ-5D | At 5 days
  Quality of life measured by EQ-5D (European Quality of Life-5 Dimensions) at POD5
EQ-5D | At 14 days
  Quality of life measured by EQ-5D at POD14
EQ-5D | At 35 days
  Quality of life measured by EQ-5D at POD35
Fatigue score | At 5 days
  Fatigue measured FACIT-F (The Functional Assessment of Chronic Illness Therapy-Fatigue) questionnaire at POD5
Fatigue score | At 14 days
  Fatigue measured FACIT-F questionnaire at POD14
Fatigue score | At 35 days
  Fatigue measured FACIT-F questionnaire at POD35
Barthel Index | At 5 days
  Independence in daily activities measured by the Barthel questionnaire at POD 5
Barthel Index | At 14 days
  Independence in daily activities measured by the Barthel questionnaire at POD 14
Barthel Index | At 35 days
  Independence in daily activities measured by the Barthel questionnaire at POD 35
Length of hospital stay | At 3 months
  Hospitalized days
Adverse events | At 3 months
  Incidence of adverse events
Infection | At 3 months
  Incidence of postoperative infection

CONTACTS AND LOCATIONS:
Overall Officials: Weiyun Chen, MD, Principal Investigator — Peking Union Medical College Hospital; Jianxiong Shen, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Coded data is anticipated to be shared with potential collaborators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Anticipated that data from the study will become available within 5 years after publication of main data.
Access Criteria: Data would only be shared with IRB approved collaborators.

REFERENCES:
- [Background] Zhan J, Jiao Y, Chen W, Huang Y, Shen J. Effects of ferric derisomaltose on postoperative anaemia in adult spinal deformity surgery: a study protocol for a randomised controlled trial. BMJ Open. 2024 Jan 24;14(1):e080952. doi: 10.1136/bmjopen-2023-080952. PMID 38267243